CLINICAL TRIAL: NCT07109661
Title: EFFICACY OF THE RATIONAL POSITIVE PARENTING PROGRAM (rPPP) FOR DISRUPTIVE BEHAVIORS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sadia Ramzan (Other)
Responsible Party: Sponsor-Investigator, Sadia Ramzan, MS Scholar, Clinical Psychology, University of the Punjab
Organization: University of the Punjab (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. D/114/FIMS
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Disruptive Behaviors
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Participants (caregivers of children with disruptive behaviors) will be randomly assigned to either the intervention group (receiving rPPP sessions) or the waitlist control group. The intervention group will complete weekly sessions of the Rational Positive Parenting Program, while the control group will receive usual care and be offered the intervention after post-assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receiving Rational Positive Parenting Program (rPPP) throughout the study.
  Interventions: Behavioral: Rational Positive Parenting Program (rPPP)
- Waitlist Control Group (Other): Participants on waitlist control, they will receive the rPPP after post-intervention assessment.
  Interventions: Behavioral: Rational Positive Parenting Program (rPPP)

INTERVENTIONS:
Behavioral: Rational Positive Parenting Program (rPPP) — The Rational Positive Parenting Program (rPPP) is a structured cognitive-behavioral group intervention based on Rational Emotive Behavior Therapy (REBT). It comprises 8-10 weekly sessions focused on addressing irrational parenting beliefs, improving emotion regulation, and teaching positive behavior management strategies for children with disruptive behaviors. Participants in the control group will not receive the intervention during the active phase, but will be offered the rPPP after final assessment to ensure ethical treatment.

SUMMARY:
The goal of this clinical trial is to learn if the Rational Positive Parenting Program (rPPP), a group-based intervention based on Rational Emotive Behavior Therapy (REBT), can help reduce disruptive behaviors in children and improve parenting among mothers in Pakistan. The study focuses on mothers of children aged 6-12 years who show behavioral problems like aggression, defiance, and temper outbursts.

The main questions it aims to answer are:

Does the rPPP reduce disruptive behavior in children? Does it improve parents' beliefs, emotional regulation, and sense of competence? Researchers will compare a group of mothers receiving the rPPP to a wait-list control group to see if the intervention leads to positive changes in both parent and child behavior.

Participants will:

Attend weekly group sessions based on rPPP techniques. Complete assessments before and after the program using standardized tools. Be followed up to evaluate the program's effectiveness in improving parenting and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For Mothers

  1. Mothers with the age range between 30 and 45 years.
  2. Mothers who score high on the PAS and P RIBS will be included in the study.
  3. Mothers willing and available to attend group-based rPPP sessions throughout the intervention period.

For Children

1. Children between 6 and 12 years of age.
2. Children who score 131 or above on the Intensity Scale or 15 or above on the Problem Scale of the Eyberg Child Behavior Inventory (ECBI).

Exclusion Criteria:

* For Mothers

  1. Mothers with Psychological illness (screening questions will be included in the demographic section),
  2. Mothers enrolled in any other parenting or psychological intervention programs. For Children

  <!-- -->

  1. Children with comorbid neurodevelopmental disorders (e.g., autism, ADHD) (screening questions will be included in the demographic section)

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory - ECBI | Baseline and after 8 weeks of intervention
Parenting Sense of Competence Scale - PSCS | Baseline and after 8 weeks of intervention
Parent Rational and Irrational Belief Scale - PRIBS | Baseline and after 8 weeks of intervention
Parent Anger Scale - PAS | Baseline and after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hira Liaqat Supervisor, Principal Investigator — Centre for Clinical Psychology, University of the Punjab
Locations (1):
- Centre for Clinical Psychology, University of the Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided